CLINICAL TRIAL: NCT02183051
Title: A Short Term Double-blind Trial to Compare the the Analgesic Efficacy and Tolerability of Meloxicam 15 mg, 7.5 mg, 3.75 mg and 1.875 mg Oral (Quick Tablet) Versus Placebo and Ibuprofen 400 mg and 200 mg Oral in the Treatment of Pain After Surgery of the Third Molar
Brief Title: Study to Compare the the Analgesic Efficacy and Tolerability of Meloxicam Versus Placebo and Ibuprofen in the Treatment of Pain After Surgery of the Third Molar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107.197
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Meloxicam; Ibuprofen

ARMS (7):
- Meloxicam 15 mg (Experimental)
  Interventions: Drug: Placebo; Drug: Meloxicam 15 mg
- Meloxicam 7.5 mg (Experimental)
  Interventions: Drug: Meloxicam 7.5 mg; Drug: Placebo
- Meloxicam 3.75 mg (Experimental)
  Interventions: Drug: Meloxicam 3.75 mg; Drug: Placebo
- Meloxicam 1.875 mg (Experimental)
  Interventions: Drug: Meloxicam 1.875 mg; Drug: Placebo
- Ibuprofen 400 mg (Active Comparator)
  Interventions: Drug: Placebo; Drug: Ibuprofen 400 mg
- Ibuprofen 200 mg (Active Comparator)
  Interventions: Drug: Ibuprofen 200 mg; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meloxicam 7.5 mg
  Arms: Meloxicam 7.5 mg
Drug: Meloxicam 3.75 mg
  Arms: Meloxicam 3.75 mg
Drug: Meloxicam 1.875 mg
  Arms: Meloxicam 1.875 mg
Drug: Ibuprofen 200 mg
  Arms: Ibuprofen 200 mg
Drug: Placebo
Drug: Meloxicam 15 mg
  Arms: Meloxicam 15 mg
Drug: Ibuprofen 400 mg
  Arms: Ibuprofen 400 mg

SUMMARY:
To assess the analgesic efficacy and tolerability of meloxicam 15 mg, 7.5 mg, 3.75 mg and 1.875 mg oral (rapid release tablet) compared with placebo and ibuprofen 400 mg and 200 mg administered in a single dose, over an observation period of 6 hours in the treatment of pain after surgery of the third molar.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above
* Patients undergoing removal of one impacted mandibular third molar under local anesthesia. (Short duration anaesthetics will be allowed, i.e. mepivacaine 3% in Italy and Spain and xylocaine in USA, both without vasoconstrictors) Only patients with type of inclusion II to IV have to be included (type II, molar in the submucosa; type III, molar partially included in the bone; type IV, molar fully included in the bone)
* Assessment of pain must be at least 50 mm on a 100 mm visual analogue scale (VAS)
* Patient informed consent in accordance with local legislation.

Exclusion Criteria:

* Type I of inclusion (molar partially or totally erupted)
* Known or suspected hypersensitivity to trial drug or their excipients, analgesics, antipyretics or nonsteroidal antiinflammatory drug (NSAIDs)
* Any clinical evidence of active peptic ulceration during the last six month
* Recurrent ulcers
* Pregnancy or breast feeding
* Asthma, nasal polyps, angioneurotic oedema or urticaria following the administration of aspirin or NSAIDs
* Concomitant treatment with anti-coagulants (including heparin), lithium
* Concomitant administration of other anti inflammatory or analgesic agents
* Administration of any drug with analgesic properties in the 24 h previous to the administration of the study drug, except the local anesthetic for the surgery
* Administration of any antibiotics
* Significant perioperative complication judged by the oral surgeon
* Clinical evidence of or known severe cardiac, hepatic, renal, metabolic, hematological disease (including bleeding disorders), mental disturbance, ulcerative colitis
* Any other disease that could interfere with the evaluation of efficacy and safety
* Participation in another clinical trial during this study or during the previous month
* Previous participation in this trial
* Patient unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 1998-04; Primary Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Assessment of pain intensity differences (PID) on a visual analogue scale (VAS, 100 mm) from one hour onwards | 60, 90, 120, 180, 240, 300 and 360 minutes after drug administration

SECONDARY OUTCOMES:
Assessment of PID on a VAS | Up to 360 minutes after drug administration
Sum of pain intensity differences (SPID) | Up to 360 minutes after drug administration
Number of patients with pain decrease >=50% | Up to 360 minutes after drug administration
Assessment of maximum pain decrease on a VAS | Up to 360 minutes after drug administration
Number of withdrawals due to safety reasons | Up to 7 days after drug administration
Number, nature and severity of adverse events | Up to 7 days after drug administration
Total pain relief (TOTPAR) assessed by patient (Area under the pain relief-by time curve) | Up to 360 minutes after drug administration
Assessment of onset of analgesic action | Up to 2 hours after surgery
Final assessment of efficacy by patient on a 4-point verbal rating scale (VRS) | 6 hours after drug administration
Final assessment of efficacy by investigator on a 4-point VRS | 2 hours after drug administration
Change from baseline in laboratory values | Baseline, up to 7 days after drug administration
Assessment of the progress of healing of the extraction site | 3-7 days after drug administration
Patient's assessment of overall tolerability on a 4-point rating scale | Day 7 after drug administration
Investigator's assessment of overall tolerability on a 4-point rating scale | Day 7 after drug administration
Pain relief assessed by patient on a 5-point VRS | Up to 360 minutesafter drug administration
Number of withdrawals due to inadequate efficacy | Up to 7 days after drug administration